CLINICAL TRIAL: NCT06184893
Title: Multi-centric Prospective and Observational Study of Prevalence and Incidence of Interstitial Lung Diseases in Patients With Rheumatoid Arthritis
Brief Title: Rheumatoid Arthritis-associated Interstitial Lung Disease Definition
Acronym: RAID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Denis Anna, Medical doctor, Centre Hospitalier Universitaire de Liege
Other Study IDs: 2022/52
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Rheumatoid Arthritis-Associated Interstitial Lung Disease
Keywords: rheumatoid arthritis; rheumatoid arthritis-associated interstitial lung disease; interstitial lung disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- General cohort
- RAIDbio: Sub-cohort studying biomarkers: volatile organic compounds, induced sputum and blood biomarkers
- RAIDomix: Sub-cohort studying radiomic patterns (based on high resolution computed tomography of the chest)

SUMMARY:
This is a prospective multicenter study in southern Belgium to determine the prevalence and incidence of interstitial lung disease in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This is a prospective multi-centric longitudinal study of the prevalence and incidence of pulmonary diseases in patients with RA.

During one year, patients with a RA diagnosis (according to the criteria of the American Society of Rheumatology) in the south of Belgium will be enrolled on a voluntary basis. If available, data including quality of life and symptoms questionnaires, medical examinations, 6-minute walk-tests, pulmonary function tests and chest CT will be collected during two years.

Furthermore, patients could be included (if available data) in two additional sub-cohorts:

* "RAIDbio" sub-cohort studying biomarkers: volatile organic compounds, induced sputum and blood biomarkers;
* "RAIDomix" sub-cohort studying radiomic patterns (based on high resolution computed tomography of the chest).

Due to a non-specific and poor clinical expression at beginning, there is currently an under-diagnosis of rheumatoid arthritis associated-interstitial lung disease (RA-ILD) at an early stage and we assume that an annual pneumological follow-up, search of early biomarkers and a radiomic approach of RA patients will overcome this issue. This should lead to a better follow-up and management (including the use of anti-fibrotic therapies in the future) of these patients and ultimately to a decrease in morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis according to the criteria of the American Society of Rheumatology
* Age > 18 years
* Willing to participate in the study and sign the informed consent form (ICF) of participants or their legal authorized representative
* RAIDbio subcohort : available data for one of the following analysis of biomarkers: volatile organic compounds, induced sputum or blood markers
* RAIDomix : available data for high resolution computed tomography of the chest

Exclusion Criteria: none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis visiting their rheumatologist in South of Belgium and willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence | 2-5 years
  To determine real-life prevalence and incidence of lung diseases in all patients with RA in South of Belgium

SECONDARY OUTCOMES:
Early diagnosis | 2-5 years
  To diagnose RA-ILD at an earlier stage
Morbidty/mortality | 2-5 years
  To decrease the morbidity and mortality associated with RA-ILD
Biomarkers | 2-5 years
  To identify specific early biomarkers of RA-ILD
Radiomics | 2-5 years
  To evaluate the prognosis value of radiomics approach in RA-ILD

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Liege, Liège, Belgium